CLINICAL TRIAL: NCT06497998
Title: Use of the EGG Sensor to Characterize Human Oocytes in IVF With ICSI
Brief Title: EGG Sensor for Oocyte Characterization
Acronym: EGG_SENSOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023/776
Record Dates: First submitted 2024-06-27; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGG sensor (Experimental): Mechanical characterization is performed using a glass indenter that applies a load to the oocyte.
  The indenter is a sterile, single-use, blunt-edged glass cylinder with a flat support end featuring a small foam formation, approximately the diameter of a micropipette.
  Except for the mechanical characterization, all oocytes are managed similarly according to validated procedures: in the same location, under the same metrological constraints (temperature and pH (potential of hydrogen) monitoring), and are handled by the same competent ART personnel.
  Interventions: Device: Mechanical characterization
- Standard (No Intervention): Usual ICSI procedures

INTERVENTIONS:
Device: Mechanical characterization — The oocyte is placed in a culture dish with IVF culture medium. This procedure is similar to that used in the ICSI procedure, except that the injection pipette is replaced by a glass indenter. The indenter (sterile, single-use, blunt-edged glass cylinder, L:16mm, ø:0.85mm, mass:8mg) is completely decoupled from the micromanipulation and microinjection platform and driven by the principle of a magnetic spring with negative stiffness.
  The oocyte is immobilized using a restraining pipette to prevent unwanted movement during measurement.
  The main objective is to investigate the prognostic value of parameters derived from kinetic measurements of microforces on mature human oocytes in the context of IVF with ICSI.
  On each oocyte the mechanical testing is divided in 4 successive loading unloading phase to measure:
  * global elasticity of the oocyte.
  * global viscosity behaviour of the oocyte.
  * local elasticity of the oocyte.
  * local viscosity behaviour of the pellucid membrane.
  Arms: EGG sensor

SUMMARY:
While intracytoplasmic sperm injection (ICSI) has made significant progress in the treatment of male infertility, the cumulative delivery rate is less than 30%, and birth is sometimes only achieved after several transfers. This success rate, combined with the possibility of repeated transfer failures, causes great distress, impacting couples' personal, social, and professional lives. These failures also have a significant economic impact on society and assisted reproductive technologies (ART) laboratories, including costs related to personnel, consumables, and cryopreservation activities.

Among the factors influencing the success of ICSI, the quality of the oocyte is paramount. Identifying mature oocytes with high birth potential is therefore a crucial step in any attempt.

At present, oocyte selection is mainly based on subjective visual morphological criteria, primarily limited to the stage of meiotic maturation. Various objective selection criteria are currently being tested, such as markers in follicular fluid or the transcriptome of cumulus and granulosa cells.

Mechanical oocyte characterization is another objective approach to assessing oocyte quality. EGG Sensor is a reliable, cost-effective platform that measures forces ranging from a few nanonewtons to a few micronewtons in a liquid medium on living cells. It enables the characterization of the mechanical behavior of oocytes (kinetic measurements of forces resulting from EGG sensor action).

The EGG sensor has been evaluated, enabling the EGG platform to be duplicated at the ART center of the Besançon University Hospital, making measurement and calibration more reliable, and allowing for the characterization of a series of oocytes excluded from the ICSI procedure.

The preclinical stages in the development of the EGG sensor have thus been validated. The next stage of development is to validate the device in an operational environment. The aim of this pilot study is to evaluate the mechanical qualification of oocytes by the EGG sensor in real-life conditions during an ICSI-type ART attempt.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 43 years old.
* Candidates for in vitro fertilization with ICSI treatment
* Male infertility (with the exception of testicular sperm extraction (TESA or MESA), donation of sperm and oocytes).
* Normal mobility and morphology of sperm selected for ICSI.
* Agreement given by the multidisciplinary team of the ART center (patients considered to have a "good prognosis" at the conclusion of the meeting, with normal ovarian reserve (follicular count between 15 and 25), and candidates for single embryo transfer.
* Consenting to the EGG sensor examination of 50% of mature oocytes collected.
* Signed informed consent.
* Affiliated to the French social security system (including CMU).

Exclusion Criteria:

* age < 18 years
* age > 43 years
* Infertility of female origin (severe endometriosis, genetic origin, uterine malformations that may interfere with implantation, etc.).
* Opposition of the multidisciplinary team of the ART center and/or patients with poor or average prognosis at the conclusion of the multidisciplinary ART meeting.
* Person under legal protection and/or unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator
* Subject without health insurance
* Subject is in the exclusion period of another study or listed in the "volunteers' registry

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Differences in the global elasticity of the oocyte depending on whether or not it results in a live birth. | 36 months
  Global elasticity obtained from a loading and unloading test at constant speed using a large flat shape to compress it. The output is a curve related to the force applied to the oocyte versus the indentation depth. This curve is representative of the global oocyte elasticity.
Differences in the global viscosity behaviour of the oocyte depending on whether or not it results in a live birth | 36 months
  Global viscosity behaviour obtained from a loading test at constant speed followed by keeping the indentation depth. In this test, we are also using the large flat shape of indenter tip.The output is a curve related to the force applied to the oocyte versus time that quantify the global relaxation phenomenon of the oocyte.
Differences in the local elasticity of the oocyte depending on whether or not it results in a live birth | 36 months
  Local elasticity obtained from a loading and unloading test at constant speed using a sharp shape in order to specifically characterize pellucid membrane. The output is a curve related to the force applied to the oocyte versus the indentation depth. This curve is representative of the pellucide membrane elasticity.
Differences in the local viscosity of the pellucid membrane depending on whether or not it results in a live birth | 36 months
  Local viscosity behaviour of the pellucid membrane obtained from a loading test at constant speed followed by keeping the indentation depth. In this test, we are also using the sharp shape of indenter tip.The output is a curve related to the force applied to the oocyte versus time that mainly quantify the local relaxation phenomenon of the pellucid membrane.

SECONDARY OUTCOMES:
Differences in the mechanical characterization of an oocyte depending on whether or not it results in an early or late miscarriage. | 36 months
Differences in the mechanical characterization of an oocyte depending on whether or not it results in a clinical pregnancy. | 36 months
Differences in the mechanical characterization of an oocyte depending on whether or not it results in a biochemical pregnancy. | 36 months
Morphological characterization of mature oocytes (included in the ICSI procedure) and of abnormal or immature oocytes (excluded from the ICSI procedure). | On the day the IVF with ICSI is performed
Mechanical characterization of abnormal or immature oocytes (excluded from the ICSI procedure) from the same cohort. | On the day the IVF with ICSI is performed
Associations between oocytes' mechanical characteristics and patients' clinical and demographic characteristics. | 36 months
  Patients' clinical and demographic data include age, medical history (smoking, fertility status), the number of obtained oocytes..
Biochemical pregnancy rates | 36 months
Early and late miscarriages rates | 36 months
Clinical pregnancy rates | 36 months
Live births rates | 36 months

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date
Access Criteria: Researchers who submit a methodologically sound proposal approved by our research team